CLINICAL TRIAL: NCT04746144
Title: Return to Physical Activities and Aerobic Fitness After Total Knee Arthroplasty in Younger Patients
Brief Title: Return Physical Activities After Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Cincinnati Sportsmedicine Research and Education Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: TKRActivity13-15
Record Dates: First submitted 2021-02-02; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Total Knee Arthroplasty
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Total knee arthroplasty

SUMMARY:
The ability to resume physical activities, aerobic fitness and a healthy lifestyle without symptoms after total knee arthroplasty (TKA) remains unclear because studies show high rates of patient dissatisfaction. The aim of this study was to evaluate whether an individualized goal-centered rehabilitation protocol leads to high patient-reported physical activities and satisfaction after TKA.

DETAILED DESCRIPTION:
A prospective study was conducted in patients who underwent primary TKA (Journey II, Smith & Nephew) from the same surgeon from July 1, 2013 to December 31, 2015. Patients completed patient-reported outcome measures (PROMs) before the operation and then at 1, 2, and 4 years postoperatively.These included the Knee Injury and Osteoarthritis Outcome Joint Replacement Survey (KOOS JR) 7-item score; questions from the Cincinnati Knee Rating System related to the overall knee condition, pain, and swelling; selected questions from the Veterans RAND 12-Item Health Survey; questions about general fitness level; and questions regarding patient expectations before and after surgery. Patients were asked to list all physical, recreational, and work activities they participated in after surgery. An experienced research associate interviewed the patients postoperatively, with data reduction and patient ratings blinded to the treating surgeon and therapist.

ELIGIBILITY:
Inclusion Criteria:

* Age < 70 years
* Patient goals to return to recreational and occupational activities
* Agree to participate in a postoperative rehabilitation and home exercise program

Exclusion Criteria:

* Osteoarthritis in other joints
* Co-morbidities limiting physical activity
* Presence of a connective tissue disease
* Autoimmune disease or immune deficiency
* Age 70 years or more
* no desire to return to recreational and work activities
* Refusal to participate in rehabilitation program

Max Age: 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients were selected from the treating surgeon's patient population.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Joint Replacement Survey (KOOS) Jr 7-item score | Preoperative
  Scored on a scale of 0-100 points, where 0 = total disability and 100 = perfect knee health.
Knee Injury and Osteoarthritis Outcome Joint Replacement Survey (KOOS) Jr 7-item score | 4 years postoperative
  Scored on a scale of 0-100 points, where 0 = total disability and 100 = perfect knee health.
Documentation of sports and recreational activities | 4 years postoperative
  Patients provide a list of all sports and recreational activities they participated in after surgery. This is an open-ended question "What sports or recreational activities do you participate in on a regular basis?"

SECONDARY OUTCOMES:
Cincinnati Knee Rating Pain Score | Preoperative
  Scored on a point scale where patient selects 0, 2, 4, or 6; where 0 = severe pain constant with daily activities, 2 = moderate pain with activities of daily living, 4 = able to do activities of daily living with no pain, and 6 = no pain with recreational activities
Cincinnati Knee Rating Pain Score | 4 years postoperative
  Scored on a point scale where patient selects 0, 2, 4, or 6; where 0 = severe pain constant with daily activities, 2 = moderate pain with activities of daily living, 4 = able to do activities of daily living with no pain, and 6 = no pain with recreational activities
Cincinnati Knee Rating Patient Perception of the Overall Knee Condition Score | Preoperative
  Score for the patient rating of the overall knee condition (0-10 point scale where 0 = poor and 10 = excellent)
Cincinnati Knee Rating Patient Perception of the Overall Knee Condition Score | 4 years postoperative
  Score for the patient rating of the overall knee condition (0-10 point scale where 0 = poor and 10 = excellent)
Cincinnati Knee Rating Swelling Score | Preoperative
  Scored on a point scale where patient selects 0, 2, 4, or 6; where 0 = severe swelling constant with daily activities, 2 = moderate swelling with activities of daily living, 4 = able to do activities of daily living with no swelling, and 6 = no swelling with recreational activities
Cincinnati Knee Rating Swelling Score | 4 years postoperative
  Scored on a point scale where patient selects 0, 2, 4, or 6; where 0 = severe swelling constant with daily activities, 2 = moderate swelling with activities of daily living, 4 = able to do activities of daily living with no swelling, and 6 = no swelling with recreational activities
Aerobic fitness levels | Preoperative
  Two questions are completed:
  1. Are you able to take a brisk 20-minute walk that raises your heart rate 5 days a week?
  2. Are you able to spend 20 minutes doing vigorous aerobic activity that causes a large increase in your heart rate 3 days a week? Scale for both questions: Yes; No, because of pain in my knee; No, because of pain in another joint; No, because of other reasons
Aerobic fitness levels | 4 years postoperative
  Two questions are completed:
  1. Are you able to take a brisk 20-minute walk that raises your heart rate 5 days a week?
  2. Are you able to spend 20 minutes doing vigorous aerobic activity that causes a large increase in your heart rate 3 days a week? Scale for both questions: Yes; No, because of pain in my knee; No, because of pain in another joint; No, because of other reasons
Work Status | Preoperative
  Single question: Are you able to work:
  Patients select: Yes, with no limitations; Yes, with limitations; No, Retired or does not apply
Work Status | 4 years postoperative
  Single question: Are you able to work:
  Patients select: Yes, with no limitations; Yes, with limitations; No, Retired or does not apply
Patient Expectations After Surgery | 4 years postoperative
  4 questions:
  1. My expectations for being able to do my normal activities of daily living after the knee surgery were:
  2. My expectations for being able to do my leisure, recreational or sports activities after the knee surgery were:
     Scale for first 2 questions: Too low, I'm a lot better than I thought; Too low, I'm somewhat better than I thought; Just right, my expectations were met; Too high, I'm somewhat worse than I thought; Too high, I'm a lot worse than I thought.
  3. Was your surgery worthwhile; are you glad you underwent the procedure? Scale: Yes, definitely; Yes, probably; No, probably; No, definitely
  4. Compare the overall condition of your knee now to what it was before your surgery.
  Scale: Great deal better, Somewhat better, The same, Somewhat worse, Great deal worse
Patient Expectations Before Surgery | Preoperative
  2 questions:
  1. I expect that, after my knee surgery, activities such as walking, stairs, and kneeling to be:
  2. I expect that, after my knee surgery, recreational activities such as bicycling, hiking, golf, light tennis, to be:
  Scale for both questions: Fully normal with no limitation; Almost normal with some limitations; Improved, but may have some problems; Improved, but may have bothersome problems; Not possible or not interested in recreational activities

CONTACTS AND LOCATIONS:
Overall Officials: Frank R Noyes, MD, Principal Investigator — Cincinnati Sportsmedicine and Orthopaedic Center
Locations (1):
- Cincinnati Sportsmedicine and Orthopaedic Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No